CLINICAL TRIAL: NCT03911154
Title: Evaluation of SmartSleep Technology for Improving the Efficiency and Restorative Quality of Sleep in Healthy Adults in Order to Mitigate Cognitive Performance Deficits Due to Sleep Restriction and Emergency Awakenings
Brief Title: Evaluation of SmartSleep Technology for Improving the Efficiency and Restorative Quality of Sleep in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Aeronautics and Space Administration (NASA) (U.S. Federal Agency); Philips Healthcare (Industry); University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: NNX16AO69A/T0408
Record Dates: First submitted 2019-04-04; First posted 2019-04-10 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-09

CONDITIONS: Sleep
Keywords: Sleep; Sleep restriction; Cognitive performance

STUDY DESIGN:
Intervention Model Description: This study uses within subject randomization. Each subject will receive all of the 4 sleep conditions in a randomized order that will be unknown to the subject.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The SmartSleep device will be programmed by investigators not involved in study execution. Subjects will wear the SmartSleep device each night and will be unaware of the order of stimulation modalities. In addition, both study personnel and those assessing outcomes will not be aware of the order of stimulation modalities.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- SmartSleep Continuous Fixed Interval modality (Experimental): This study uses within subject comparison. For each subject, the order of 3 SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 3 stimulation modalities and a SHAM condition.
  This study arm tests the SmartSleep Continuous Fixed Interval stimulation modality during sleep relative to the SHAM condition. The Continuous Fixed Interval is the delivery of auditory tones a 1 Hz inter-tone interval stimulation.
  Interventions: Device: Philips SmartSleep Technology--Continuous Fixed Interval modality; Device: Philips SmartSleep Technology--Block modality; Device: Philips SmartSleep Technology--In-Phase Adjustable modality
- SmartSleep Block modality (Experimental): This study uses within subject comparison. For each subject, the order of 3 SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 3 stimulation modalities and a SHAM condition.
  This study arm tests the SmartSleep Block stimulation modality during sleep relative to the SHAM condition. The Block is the delivery of auditory tones for 5 seconds on versus 5 seconds off.
  Interventions: Device: Philips SmartSleep Technology--Continuous Fixed Interval modality; Device: Philips SmartSleep Technology--Block modality; Device: Philips SmartSleep Technology--In-Phase Adjustable modality
- SmartSleep In-Phase Adjustable modality (Experimental): This study uses within subject comparison. For each subject, the order of 3 SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 3 stimulation modalities and a SHAM condition.
  This study arm tests the SmartSleep In-Phase Adjustable stimulation modality during sleep relative to the SHAM condition. The In-Phase Adjustable is the constant stimulation with auditory tones delivered during each upstate of the slow wave.
  Interventions: Device: Philips SmartSleep Technology--Continuous Fixed Interval modality; Device: Philips SmartSleep Technology--Block modality; Device: Philips SmartSleep Technology--In-Phase Adjustable modality
- SHAM condition (Sham Comparator): This study uses within subject comparison. For each subject, the order of 3 SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 3 stimulation modalities and a SHAM condition.
  This study arm is the SHAM condition, during which participants wore the SmartSleep device, however no auditory tones were delivered.
  Interventions: Device: Philips SmartSleep Technology--Continuous Fixed Interval modality; Device: Philips SmartSleep Technology--Block modality; Device: Philips SmartSleep Technology--In-Phase Adjustable modality

INTERVENTIONS:
Device: Philips SmartSleep Technology--Continuous Fixed Interval modality — During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval
  2. Block
  3. In-Phase Adjustable
  4. Sham: No auditory stimulation while wearing the SmartSleep headband
Device: Philips SmartSleep Technology--Block modality — During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval
  2. Block
  3. In-Phase Adjustable
  4. Sham: No auditory stimulation while wearing the SmartSleep headband
Device: Philips SmartSleep Technology--In-Phase Adjustable modality — During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval
  2. Block
  3. In-Phase Adjustable
  4. Sham: No auditory stimulation while wearing the SmartSleep headband

SUMMARY:
This study aims to assess whether slow wave sleep enhancement using SmartSleep technology benefits daytime cognitive performance during periods of chronic sleep restriction.

DETAILED DESCRIPTION:
Adequate healthy sleep is essential in spaceflight to ensure that astronauts maintain a high level of cognitive performance capability and do so without undue stress. There is a need for a technology that can improve sleep quality in space and biologically maximize the performance benefits of limited sleep duration, without unduly affecting the ability of astronauts to awaken abruptly and respond to an in-flight emergency. Sleep slow waves support system and synaptic consolidation by promoting specific patterns of neuromodulatory and electric activities, and subjective sleep quality is related to the size and number of slow waves that occur nightly.

This study will use SmartSleep (Philips) technology to determine what effect the device has on daytime cognitive performance after emergent awakenings from sleep in a chronic sleep restriction paradigm. The SmartSleep technology uses two small sensors in the headband to continuously detect the brain's slow wave sleep (delta/theta frequency) in real time, and a closed-loop algorithm customizes the timing and volume of tones to optimize the sleep pattern. Thus, the device uses "quiet audio tones" (sub-awareness) to increase slow waves, which can enhance sleep quality/depth, thereby enhancing subsequent waking cognitive performance without the unwanted sedating effects of medications on cognitive functions during emergency awakenings.

Subjects will be in the laboratory for 7 days/6 nights. Night 1 will be an adaptation night with 8-hours time in bed. Nights 2-5 will consist of 5 hours time in bed, followed by night 6 of a recovery 10 hours time in bed. During nights 2-5, subjects will receive one of four stimulation modalities using the SmartSleep wearable device. Subjects will receive all four modalities in a randomized order:

1. Continuous Fixed Interval
2. Block
3. In-Phase Adjustable
4. Sham: No auditory stimulation while wearing the SmartSleep headband

Cognitive performance testing and self-report surveys will be completed on a daily basis. A total of 12 healthy astronaut-like adults will be studied. Subjects will complete the 7-day study in groups of 4.

ELIGIBILITY:
Inclusion Criteria:

* Bachelor's degree or Master's degree (or the equivalent in work experience) in a relevant field, and/or military service.
* Free of psychological/psychiatric conditions that preclude participation.
* BMI < 35.
* Self-reported regular sleep schedule; able to maintain their sleep schedule during the course of the study.
* Self-reported sleep duration of 6-8.5 hrs per night (verified by 6 work days of ambulatory sleep monitoring with wrist actigraphy and daily logs).
* Ability to read/write English.

Exclusion Criteria:

* History of neurological, psychiatric, or other medical condition that excludes participation.
* Current mania or psychosis.
* Current depression as determined by the Beck Depression Inventory (Beck, 1996).
* Alcohol or drug abuse in the past year based upon history and urine toxicology screen.
* Excessive alcohol intake (≥ 21 drinks per week) or binge alcohol consumption (> 5 drinks per day).
* Excessive caffeine consumption (> 650mg/day combining all caffeinated drinks regularly absorbed during the day).
* Current smoker/tobacco user, or using nicotine replacement therapy. Those that have been nicotine-free for 30 days will be included.
* Acute, chronic, or debilitating medical conditions, major Axis I psychiatric illness based on history, physical exam, blood and urine chemistries, and CBC.
* Individuals who self-report a history of recurrent seizures or epilepsy or have a history of medical conditions that could increase the chance of seizures (e.g. stroke, aneurysm, brain surgery, structural brain lesion).
* Cardiovascular, neurological, gastrointestinal, or musculoskeletal problems that exclude participation.
* Major controlled or uncontrolled medical condition such as congestive heart failure, neuromuscular disease, renal failure, cancer, COPD, respiratory failure or insufficiency, or patients requiring oxygen therapy (as determined by self-report).
* Currently working night, swing, split or rotating shift.
* Current use or use of within the past month of a prescription or over-the-counter sleep medication or stimulant; use of psychoactive medication (based on self-report and review with a study clinician).
* Pregnant or currently breast feeding
* Prior history or diagnosis of any sleep disorder
* High Risk of OSA based on STOP-BANG Questionnaire ("yes" on at least 4 of 8 questions)
* High Risk of Restless Legs Syndrome (RLS) based on Cambridge-Hopkins Screening questionnaire
* High Risk of Insomnia based on Insomnia Severity Index (score of 22 or higher)
* Individuals who self-report severe contact dermatitis or allergy to silicone, nickel or silver.
* Individuals who self-report moderate hearing loss.
* Inability to achieve appropriate headband fit.
* Planned travel across more than one time zone one month prior to and/or during the anticipated period of the study with SmartSleeps device use.
* Intentional naps during the week.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There are no pre-assignment events to report.
Groups:
- SmartSleep Stimulus Modality: This study uses within subject comparison. For each subject, the order of SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 4 stimulation modalities.
  Please refer to the attached study design and protocol for additional information.
  Philips SmartSleep Technology: During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval: 1 Hz inter-tone interval stimulation
  2. Block: 5 seconds on versus 5 seconds off
  3. In-Phase Adjustable: constant stimulation with tones to be delivered during each upstate of the slow wave
  4. Sham: No auditory stimulation while wearing the SmartSleep headband
Period: Overall Study
Arm/Group | SmartSleep Stimulus Modality
Started | 9
Continuous Fixed Interval (Each participant will receive the SmartSleep Continuous fixed interval modality during one night of sleep restriction) | 9
Block (Each participant will receive the SmartSleep Block modality during one night of sleep restriction) | 9
In-Phase Adjustable (Each participant will receive the SmartSleep In-Phase Adjustable modality during one night of sleep restriction) | 9
SHAM (Each participant will receive the SmartSleep SHAM modality during one night of sleep restriction) | 9
Completed | 8
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population only includes participants who completed the study. A total of N=9 participants initiated the study, however one participant withdrew from the study, and therefore, the baseline analysis includes only participants who completed the study.
Groups:
- SmartSleep Modality Assignment: This study uses within subject comparison. For each subject, the order of SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 4 stimulation modalities.
  Philips SmartSleep Technology: During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval
  2. Block
  3. In-Phase Adjustable
  4. Sham: No auditory stimulation while wearing the SmartSleep headband
Arm/Group | SmartSleep Modality Assignment
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8
PVT lapses of attention [Mean (Standard Deviation); unit: PVT lapses] — This study-specific baseline measure is the average number of PVT lapses, a measure of vigilant attention, on the baseline day following the 8-hour adaptation night of the study (night 1). The number of lapses of attention were measured by the PVT-B and a lapse of attention was defined as a response time >355 ms.
  PVT lapses | 2.44 (4.98)

OUTCOME MEASURES:

1. Primary Outcome: Psychomotor Vigilance Test-Brief (PVT-B)
Description: The PVT is a simple reaction time test that requires participants to react, as quickly as possible, by pressing a response key as soon as a rolling number counter presented in a box in the center of the computer screen appears. The PVT is a validated and widely-used measure of vigilant attention that is sensitive to the effects of sleep loss. The primary outcome was the number of PVT lapses. The minimum number of PVT lapses is "0" and there is no maximum number of lapses, which are defined as response times >355 ms. More PVT lapses indicates worse performance.
Time Frame: Days 3-6
Measure: Mean (Standard Deviation); unit: PVT lapses
Arm/Group | SmartSleep Modality Assignment
Number analyzed (Participants) | 8
PVT lapses
  Continuous Fixed Interval | 3.59 (8.18)
  Block | 4.61 (10.98)
  In-Phase Adjustable | 5.55 (13.02)
  Sham | 3.95 (9.11)
Statistical Analysis 1: Comparison: SmartSleep Modality Assignment; Number of lapses of attention were averaged across assessments within each day and the statistical analysis adjusted for baseline; Test type: Other — We used linear mixed effect models (in SAS version 9.4, SAS Institute, Cary, NC) with random subject intercept to account for the clustered nature of the data. The model included factors for stimulus modality (4 levels), sleep restriction night (4 levels), and their interaction; p = 0.36, Mixed Models Analysis; Mean Difference (Net) = 0.329, 95% CI 2-sided [-0.403 to 1.060], Standard Error of Mean 0.353
Statistical Analysis 2: Comparison: SmartSleep Modality Assignment; Number of lapses of attention upon emergent awakening; Test type: Other — Linear mixed effects model with a random subject intercept; p = 0.49, Mixed Models Analysis; Mean Difference (Net) = -0.307, 95% CI 2-sided [-1.222 to 0.608], Standard Error of Mean 0.441

2. Primary Outcome: Slow-wave Activity
Description: Total delta power measured during sleep
Time Frame: Days 3-6
Measure: Mean (Standard Deviation); unit: microvolts^2
Arm/Group | SmartSleep Modality Assignment
Number analyzed (Participants) | 8
microvolts^2
  Continuous Fixed Interval | 943.13 (311.20)
  Block | 1006.00 (421.50)
  In-Phase Adjustable | 972.63 (485.36)
  SHAM | 822.38 (370.59)
Statistical Analysis 1: Comparison: SmartSleep Modality Assignment; Test type: Other — Linear mixed effects model with a random subject intercept; p = 0.87, Mixed Models Analysis; Mean Difference (Net) = 0.455, 95% CI 2-sided [-5.400 to 6.310], Standard Error of Mean 2.797

3. Secondary Outcome: Digit Symbol Substitution Test (DSST)
Description: The Digit Symbol Substitution Test (DSST) is a widely used measure of cognitive throughput and cognitive instability that is sensitive to the effects of sleep loss. The DSST was adapted from the Wechsler Adult Intelligence Scale. Participants are shown an array of symbols and with corresponding numbers on a keyboard. They are then presented the symbols one at a time in random order and must respond with the correct corresponding number as quickly as possible. The primary outcome was number correct and given the established practice effects on the DSST, this measure was corrected for practice effects. The DSST has a minimum of "0" correct responses and does not have a maximum; a higher number on the DSST represents better performance.
Time Frame: Days 3-6
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | SmartSleep Modality Assignment
Number analyzed (Participants) | 8
Correct responses
  Continuous Fixed Interval | 61.02 (11.72)
  Block | 61.73 (11.05)
  In-Phase Adjustable | 58.55 (17.68)
  Sham | 61.01 (12.41)
Statistical Analysis 1: Comparison: SmartSleep Modality Assignment; Number correct on the DSST was averaged across DSST administrations within each day and was adjusted for baseline performance; Test type: Other — Linear mixed effects model with a random subject intercept; p = 0.89, Mixed Models Analysis; Mean Difference (Net) = -0.112, 95% CI 2-sided [-1.767 to 1.543], Standard Error of Mean 0.798

4. Secondary Outcome: Descending Subtraction Task (DST)
Description: The Descending Subtraction Test (DST) is a measure of working memory that is sensitive to the effects of sleep loss. The DST requires participants to mentally subtract numbers in a sequential fashion as quickly as possible. For example, if the starting number is 987, the participant subtracts nine from 987, with the difference being 978, the participant then subtracts eight from 978, and so on subtracting by seven, six, five, four, three, two, and one, from each difference at which point, and the participant then recycles the subtraction sequence beginning at nine again. The DST has a minimum of "0" correct responses and does not have a maximum; a higher number on the DST represents better performance. The primary outcome on the DST was Number correct.
Time Frame: Days 3-6
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | SmartSleep Modality Assignment
Number analyzed (Participants) | 8
Correct responses
  Continuous Fixed Interval | 18.52 (10.18)
  Block | 19.33 (9.73)
  In-Phase Adjustable | 20.04 (10.97)
  Sham | 18.84 (9.41)
Statistical Analysis 1: Comparison: SmartSleep Modality Assignment; Number correct on the DST was averaged across DST administrations within each day and adjusted for baseline; Test type: Other — Linear mixed effects model with a random subject intercept; p = 0.76, Mixed Models Analysis; Mean Difference (Net) = -0.121, 95% CI 2-sided [-0.919 to 0.678], Standard Error of Mean 0.381

5. Secondary Outcome: Robotic On-Board Trainer (ROBoT) Task
Description: The Robotic On-Board Trainer (ROBoT) task is NASA's platform for training astronauts to perform docking and grappling maneuvers using the Canada Arm. The system is based on highly realistic 3D simulations of the arm and associated physics. The ROBoT system involves a left-hand translational controller (x/y/z directions) and a right-hand rotational controller (pitch/roll/yaw), plus two laptop computer screens. Key performance metrics include: (i) docking position accuracy, (ii) docking orientation accuracy, (iii) total task time, and (iv) smoothness of approach trajectory, which are aggregated to generate the primary outcome, which is the mean weighted score . The weighted score ranges from 0 to 10 and a lower score indicates better performance.
Time Frame: Days 3-6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SmartSleep Modality Assignment
Number analyzed (Participants) | 8
units on a scale
  Continuous Fixed Interval | 5.61 (2.09)
  Block | 5.70 (1.83)
  In-Phase Adjustable | 6.44 (2.14)
  Sham | 5.73 (2.38)
Statistical Analysis 1: Comparison: SmartSleep Modality Assignment; The mean weighted score on the ROBoT was adjusted for baseline; Test type: Other — Linear mixed effects model with a random subject intercept; p = 0.64, Mixed Models Analysis; Mean Difference (Net) = 0.085, 95% CI 2-sided [-0.286 to 0.456], Standard Error of Mean 0.179

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the duration of the study, which included study days 1-7
Groups:
- SmartSleep Continuous Fixed Interval Modality: This study uses within subject comparison. For each subject, the order of SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 4 stimulation modalities.
  Philips SmartSleep Technology: During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval
  2. Block
  3. In-Phase Adjustable
  4. Sham: No auditory stimulation while wearing the SmartSleep headband
  This study arm tests the SmartSleep Continuous Fixed Interval stimulation modality during sleep. The Continuous Fixed Interval is the delivery of auditory tones a 1 Hz inter-tone interval stimulation.
- SmartSleep Block Modality: This study uses within subject comparison. For each subject, the order of SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 4 stimulation modalities.
  Philips SmartSleep Technology: During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval
  2. Block
  3. In-Phase Adjustable
  4. Sham: No auditory stimulation while wearing the SmartSleep headband
  This study arm tests the SmartSleep Block stimulation modality during sleep. The Block is the delivery of auditory tones for 5 seconds on versus 5 seconds off.
- SmartSleep In-Phase Adjustable Modality: This study uses within subject comparison. For each subject, the order of SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 4 stimulation modalities.
  Philips SmartSleep Technology: During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval
  2. Block
  3. In-Phase Adjustable
  4. Sham: No auditory stimulation while wearing the SmartSleep headband
  This study arm tests the SmartSleep In-Phase Adjustable stimulation modality during sleep. The In-Phase Adjustable is the constant stimulation with auditory tones delivered during each upstate of the slow wave.
- SHAM Condition: This study uses within subject comparison. For each subject, the order of SmartSleep modalities for each of the 4 nights of sleep restriction will be randomized. All subjects will receive all 4 stimulation modalities.
  Philips SmartSleep Technology: During the 4 nights of sleep restriction (5 hours time in bed), subjects will have one of the following SmartSleep stimulation modalities each night in a randomized order. All subjects will receive all 4 stimulation modalities:
  1. Continuous Fixed Interval
  2. Block
  3. In-Phase Adjustable
  4. Sham: No auditory stimulation while wearing the SmartSleep headband
  This study arm is the SHAM condition, during which participants wore the SmartSleep device, however no auditory tones were delivered.
Arm/Group | SmartSleep Continuous Fixed Interval Modality | SmartSleep Block Modality | SmartSleep In-Phase Adjustable Modality | SHAM Condition
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8

LIMITATIONS AND CAVEATS:
The primary limitation of this study is the small sample size and given the small sample, caution in interpreting the results is warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/54/NCT03911154/Prot_SAP_ICF_001.pdf